CLINICAL TRIAL: NCT05642260
Title: The Short- and Long-term Effects of Fall Prevention Program on the Number of Falls Among Elderly Following Total Knee Replacement: a Pragmatic Single-blinded Randomized Controlled Trial.
Brief Title: Effects of Fall Prevention Program on the Number of Falls Among Elderly Following Total Knee Replacement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Health, Kuwait (Other Government)
Responsible Party: Principal Investigator, Dr. Hadeel Alsaleh, physiotherapy specialist, Ministry of Health, Kuwait
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2146/2022
Record Dates: First submitted 2022-11-29; First posted 2022-12-08 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Fall; Osteo Arthritis Knee; Total Knee Replacement
Keywords: fall; older people; fall prevention; TKR; rehabilitation

STUDY DESIGN:
Intervention Model Description: parallel group prospective (24 weeks) randomised single-blinded pragmatic controlled trial.
Who Masked: Outcomes Assessor
Masking Description: neither the participant nor the outcome assessor are aware of the groups allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Patients in the control group will receive a conventional physiotherapy treatment (guided by the post-TKR protocol followed at Al-Razi Orthopedic Hospital). The treatment will be delivered by four allocated physiotherapists,The treatment will be delivered by four allocated physiotherapists, and will consist of:
  1. Blood circulation exercise (i.e., ankle pumps)
  2. Quadriceps isometric exercises (i.e., quad sets).
  3. Knee ROM exercises (i.e., knee flexion and extension).
  4. Lower limb strengthening exercises (e.g., straight leg raising, short/ long arch exercises)
  5. Stretching exercises for the hamstring and calf muscles.
  6. Gait training (with and without the assistive device).
  7. Parallel bars exercises (e.g., standing hip abduction/adduction, knee flexion, squatting).
  8. Ascending/descending stairs.
  9. Home program.
- intervention (treatment) group (Experimental): Patients in the experimental group will receive a comprehensive fall prevention program (described below) integrated into the conventional physiotherapy treatment. The fall prevention program will consist of:
  1. Otago balance exercise for 12 weeks integrated with conventional physiotherapy treatment (described in the control group).
  2. Individualized advice on assistive device usage based on the participant's Berg Balance Score (BBS) revised at the 3 data collection timepoints.
  3. Environmental hazard checklist.
  4. Advice on getting their eyes checked and the use of appropriate footwear to ensure the elimination of other risk factors.
  5. Home program (consists of balance and strength training exercises).
  The treatment will be delivered by four allocated physiotherapists. The physiotherapists will receive an introductory/training session on the fall prevention program prior to the commencement of the trial.
  Interventions: Other: fall prevention programe

INTERVENTIONS:
Other: fall prevention programe — Patients in the experimental group will receive a comprehensive fall prevention program (guided by the post-TKR protocol followed at Al-Razi Orthopedic Hospital) into the conventional physiotherapy treatment
  Arms: intervention (treatment) group

SUMMARY:
the aim of the proposed research is to investigate the short and long-term effects of integrating a comprehensive fall prevention programme into conventional physiotherapy on the number of falls, balance, and functional ability among elderly following TKR. the investigator hypothesize that conventional physiotherapy integrated with a fall prevention program is more effective than conventional physiotherapy alone in improving balance and functional ability and preventing the occurrence of falls among elderly following TKR.

Study type: The proposed study is a parallel group prospective (24 weeks) randomised single-blinded pragmatic controlled trial.

Participants: Older adults operated for TKR at Al-Razi orthopedic hospital, who met the inclusion criteria.

DETAILED DESCRIPTION:
Falls constitute a serious and common threat to the health and well-being of older individuals, and this threat increases with aging. Falls in older individuals place a significant burden on the health care system as well as the caregivers (i.e., family). Importantly, however, many falls could be prevented.

Osteoarthritis (OA) of the knee is a common degenerative musculoskeletal condition among elderly that results in ambulatory dysfunction. This progressive degenerative disorder is usually associated with pain, muscle weakness, and poor balance, all of which are considered primary risk factors for falling among older adults. Total knee replacement (TKR) is the most replicable and effective orthopaedic procedure used to treat advanced-stage knee OA. The goal of TKR is to relieve pain, increase knee mobility, and improve functional ability and the overall quality of life. Despite the promising results of TKR surgery, it is associated with a high prevalence of falls. In this regard, falls rate have been reported to be between 6.2% and 42.6% in the first 12 months following TKR. Persistence of muscle weakness and poor balance may contribute to the high fall rate following TKR. This highlights the importance of targeting muscle strength and balance during rehabilitation, considering the short-term implications that could reflect on long-term recovery.

A substantial amount of evidence supports the use of exercise-based interventions (i.e., muscle strengthening and balance training) to prevent falls and fall-related injuries. A Cochrane systematic review by on 108 RCTs (n=23,407) provided high-certainty evidence that exercises, particularly balance and functional based-exercises, are more effective in reducing the falls rate compared to the control interventions. Moreover, exercise-based interventions have been shown to be superior to other interventions for mitigating age-related decline and reducing falls and falls-related injuries with the least harm and greatest cost-effectiveness.

Conventional physiotherapy following TKR involves, primarily, strengthening and knee range of motion exercises and gait re-education. However, there is a lack of balance training/exercises in the rehabilitation program. Given the high prevalence of falls following TKR, integrating a comprehensive fall prevention program into conventional physiotherapy may be of importance. Thus, the aim of the proposed research is to investigate the short and long-term effects of integrating a comprehensive fall prevention programme into conventional physiotherapy on the number of falls, balance, and functional ability among elderly following TKR.

ELIGIBILITY:
Inclusion Criteria:

* Female gender.
* Aged 60 years and older.
* Diagnosed with primary osteoarthritis of the knee.
* Underwent unilateral TKR.

Exclusion Criteria:

* revision TKR surgery
* history of systemic inflammatory conditions (i.e., rheumatoid arthritis, Lupus erythematosus),
* neurological disorders (i.e., multiple sclerosis, Parkinson's disease, stroke)
* lower limb surgery/trauma in the past 12 months
* have cognitive and/or vision impairments
* post-surgical complications (e.g., infection, intraoperative fracture)
* any health condition that may preclude them from undertaking physiotherapy.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female gender
Enrollment: 90 (Estimated)
Dates: Start 2023-01-08 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-09-08 (Estimated)

PRIMARY OUTCOMES:
falls rate | baseline
  The primary outcome measure in this trial will be the number of reported falls during the study period.The patients will be given a falls' diary to record the number of falls (if any), time of falling (e.g., early morning or late night), and the cause of falling (e.g., slippery floor, dizziness, tripping over).
falls rate | 12 weeks
  The primary outcome measure in this trial will be the number of reported falls during the study period.The patients will be given a falls' diary to record the number of falls (if any), time of falling (e.g., early morning or late night), and the cause of falling (e.g., slippery floor, dizziness, tripping over).
falls rate | 1 year
  The primary outcome measure in this trial will be the number of reported falls during the study period.The patients will be given a falls' diary to record the number of falls (if any), time of falling (e.g., early morning or late night), and the cause of falling (e.g., slippery floor, dizziness, tripping over).

SECONDARY OUTCOMES:
Knee range of motion (ROM) | baseline
  This will be measured using goniometer while the patient is laying in supine position with the operated knee fully extended. The patient will be requested to bend her knee 2-3 times before the actual measurements are taken. Then, the investigator will take three consecutive measurements of knee flexion range.
Knee range of motion (ROM) | 12 weeks
  This will be measured using goniometer while the patient is laying in supine position with the operated knee fully extended. The patient will be requested to bend her knee 2-3 times before the actual measurements are taken. Then, the investigator will take three consecutive measurements of knee flexion range.
Patient's satisfaction | 12 weeks
  In response to the question 'how satisfied are you with the results of physiotherapy treatment?'. Patients will be asked to grade their level of satisfaction on a 5-point Likert scale (1: not at all satisfied, 2: dissatisfied, 3: neutral, 4: satisfied, or 5: very satisfied).
Patient's satisfaction | 1 year
  In response to the question 'how satisfied are you with the results of physiotherapy treatment?'. Patients will be asked to grade their level of satisfaction on a 5-point Likert scale (1: not at all satisfied, 2: dissatisfied, 3: neutral, 4: satisfied, or 5: very satisfied).
Adherence: | 12 weeks
  1. Adherence to the prescribed home-program: Patient's adherence to the prescribed exercise/home program will be measured by a retrospective patient self-report scale, a simple method that has been implemented by other researchers to measure patient's adherence to the prescribed exercise. (Mallows et al., 2020, Bassett, 2003) In response to the question "If you have been requested by your physiotherapist to do exercises at home, please indicates the extent you have followed the instructions?", participants responded using a 5-point Likert scale ranging from 1 (not at all) to 5 (as advised).
  2. Adherence to physiotherapy attendance: The total number of treatment sessions received by the patient will be recorded by the treating physiotherapist.
Adherence: | 1 year
  1. Adherence to the prescribed home-program: Patient's adherence to the prescribed exercise/home program will be measured by a retrospective patient self-report scale, a simple method that has been implemented by other researchers to measure patient's adherence to the prescribed exercise. (Mallows et al., 2020, Bassett, 2003) In response to the question "If you have been requested by your physiotherapist to do exercises at home, please indicates the extent you have followed the instructions?", participants responded using a 5-point Likert scale ranging from 1 (not at all) to 5 (as advised).
  2. Adherence to physiotherapy attendance: The total number of treatment sessions received by the patient will be recorded by the treating physiotherapist.

OTHER OUTCOMES:
Numerical Pain Rating Scale NPRS | baseline, 12 weeks, 1 year
  The worst pain experienced in the last week will be measured using the Numerical Pain Rating Scale (NPRS). The NPRS requires the patients to rate their pain on a defined scale from 0-10 where 0 indicates no pain and 10 indicates the worst pain imaginable. Patients will be asked "Regarding your knee pain, how would you rate the worst pain that you have experienced during the last week?". A numeric change of two points on NPRS often represents a clinically important difference.
10-meter walk test | baseline, 12 weeks
  This test assesses walking speed in meters per second over a short distance. The subject walks without assistance for 10 meters (32.8 feet) and the time is measured for the intermediate 6 meters (19.7 feet) to allow for acceleration and deceleration.
Timed Up and Go test | baseline, 12 weeks
  This test measures, in seconds, the time taken by an individual to stand up from a standard armchair, walk a distance of 3 meters, turn, walk back to the chair, and sit down. The time taken to complete the task is strongly correlated to level of functional mobility, (i.e. the more time taken, the more dependent in activities of daily living).
Berg Balance Scale (BBS) | baseline, 12 weeks
  Is a 14-item scale designed to measure balance of the older adult in a clinical setting. Each item consists of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to complete. The total score equals 56. Score of < 45 indicates individuals may be at greater risk of falling (Berg et al., 1992).
30 second sit to stand: | baseline, 12weeks
  This test measures leg strength and endurance in older adults. The subject is encouraged to complete as many full stands as possible within 30 seconds without using their arms. The subject is instructed to fully sit between each stand. The score is the total number of stands within 30 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Hadeel H Alsaleh, PhD, Study Director — Ministry of Health
Locations (1):
- Alrazi orthopedic hospital, Kuwait City, Kuwait

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al-Saleh H, Merza E, Al-Adwanie B, Pearson S, Malliaras P. The short- and long-term effects of a fall prevention program on the frequency of falls following total knee replacement: A pragmatic single-blinded randomized controlled trial protocol. Contemp Clin Trials. 2025 Mar;150:107837. doi: 10.1016/j.cct.2025.107837. Epub 2025 Feb 6. PMID 39921156